CLINICAL TRIAL: NCT02436291
Title: Evaluation of the Efficacy of CURE-EX Treatment in Onychomycosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MB Mazor Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CURE-01
Record Dates: First submitted 2015-04-28; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CURE-EX device (Experimental): twice daily treatment with CURE-EX device for 24-30 weeks
  Interventions: Device: CURE-EX device

INTERVENTIONS:
Device: CURE-EX device — Treatment with CURE-EX device twice daily for 24-30 weeks.

SUMMARY:
Open label study to evaluate the efficacy of CURE-EX device in the treatment of onychomycosis.

DETAILED DESCRIPTION:
Each affected nail will be treated twice daily for 24-30 weeks. Efficacy will be evaluated by measuring the growth of healthy nail.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with clinical and mycological onychomycosis (by culture and smear).
2. Subjects did not receive topical antifungal treatment during the 14 days prior to commencing the study.
3. Subjects did not receive any systemic antifungal treatment during the 3 months prior to the start of the study.

Exclusion Criteria:

1. lunula infected with onychomycosis.
2. Pregnant or breast feeding female.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Nail cure as measured by measured by length of healthy nail of at least 5 mm | 24-30 weeks
  Cure measured by length of healthy nail of at least 5 mm
Nail cure as measured by culture and smear | 24-30 weeks
  Nail culture and smear

CONTACTS AND LOCATIONS:
Overall Officials: Avner Shemer, MD, Principal Investigator — Dermatology Clinic Natanya Israel
Locations (1):
- Lev Yasmin Clinic, Netanya, Israel